CLINICAL TRIAL: NCT02561650
Title: An Open-Label, Randomized, Single-Dose, Three-Period Crossover Study to Evaluate the Pharmacokinetics, Bioavailability, and Safety of COV155 Administered in Normal, Healthy Subjects Under Fed (High- and Low-Fat Meal) and Fasted Conditions
Brief Title: Pharmacokinetic, Bioavailability, and Safety Study of COV155 Administered in Healthy Subjects Under Fed and Fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: COV15010196
Record Dates: First submitted 2015-09-24; First posted 2015-09-28 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- COV155 (Experimental)
  Interventions: Drug: COV155

INTERVENTIONS:
Drug: COV155 — COV155 tablets

SUMMARY:
A single center, single dose, open-label, randomized, 3-period, 6-sequence, crossover study conducted in normal healthy subjects to evaluate the effect of a high- and low-fat meal on the pharmacokinetics (PK), bioavailability (BA), and safety of COV155.

ELIGIBILITY:
Inclusion Criteria:

1. Males and/or non-pregnant, non-lactating or postmenopausal females, between 18 and 55 years of age with a body mass index ≥ 19 and ≤ 30 kg/m2.
2. All subjects biologically capable of having children must agree and commit to the use acceptable method(s) of birth control.

Exclusion Criteria:

1. ECG abnormalities or lab values greater than 2 times the upper limit of normal.
2. Positive test results for human immunodeficiency virus (HIV), hepatitis B (HBsAg), or hepatitis C (IgG).
3. Positive urine test results for drugs of abuse or history of drug/alcohol abuse.
4. Use of marijuana, illicit drugs or nicotine-containing products.
5. Donated or had significant loss of whole blood.
6. Taken any prescription or nonprescription drugs, vitamins, minerals, or dietary/herbal supplements.
7. History of abdominal and/or pelvic surgery, cholecystectomy, gastric bypass or gastric band surgery, or cardiothoracic surgery.
8. History of anxiety, tension, agitation, psychiatric disorders, psychosis, or depression requiring hospitalization, psychotherapy, and/or medication.
9. History of acute or chronic gastrointestinal disease or any condition that may interfere with the absorption, distribution, metabolism or excretion of the study treatment.
10. History of seizures or diagnosis of epilepsy or other seizure disorder.
11. History or laboratory evidence of bleeding or clotting disorder or condition.
12. History or laboratory evidence of malignancy, stroke, diabetes, cardiac, renal, liver, and chronic pulmonary disease.
13. Have or have a history of hay fever or seasonal allergies requiring over-the-counter or prescription medications.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) | 48 hours
  To evaluate the effect of food on the pharmacokinetics and bioavailability of COV155 following administration of the formulation given as 2 tablets in healthy subjects under fasting and fed (high- and low-fat) conditions
Maximum observed plasma concentration (Cmax) | 48 hours
  To evaluate the effect of food on the pharmacokinetics and bioavailability of COV155 following administration of the formulation given as 2 tablets in healthy subjects under fasting and fed (high- and low-fat) conditions
Time to achieve the maximum observed plasma concentration (Tmax) | 48 hours
  To evaluate the effect of food on the pharmacokinetics and bioavailability of COV155 following administration of the formulation given as 2 tablets in healthy subjects under fasting and fed (high- and low-fat) conditions

REFERENCES:
- [Derived] Devarakonda K, Kostenbader K, Giuliani MJ, Young JL. Single-dose pharmacokinetics of 2 or 3 tablets of biphasic immediate-release/extended-release hydrocodone bitartrate/acetaminophen (MNK-155) under fed and fasted conditions: two randomized open-label trials. BMC Pharmacol Toxicol. 2015 Nov 27;16:31. doi: 10.1186/s40360-015-0032-y. PMID 26614499